CLINICAL TRIAL: NCT05362994
Title: Feasibility and Safety of Selution SLR™ Sirolimus-eluting Balloon in Patients With Distal Internal Pudendal-penile Artery Disease and Erectile Dysfunction: : PERFECT-SELUTION First-in-man (FIM)
Brief Title: Selution Sirolimus-eluting Balloon for Internal Pudendal-penile Artery Disease-related Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: M.A. Med Alliance S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202105008DIPB
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-01

CONDITIONS: Erectile Dysfunction; Peripheral Arterial Disease; Arterial Stenosis
Keywords: angioplasty; drug-coated balloon; erectile dysfunction; pelvic artery disease; peripheral artery disease; pudendal artery; penile artery
MeSH Terms: conditions — Erectile Dysfunction; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Randomization will take place before angioplasty. Patients will be randomized to either the plain old balloon (POB) group or the drug-eluting balloon (DEB) group. Three minutes after balloon predilation, the investigators will obtain an angiogram. If the residual stenosis is ≤30%, no further intervention will be performed in the plain old balloon (POB) group. While in the drug-eluting balloon (DEB) group, the investigators will perform angioplasty with the Selution SLR catheter, inflated at nominal pressure for at least 120 seconds. After dilatation of the entire target-lesion, biplane angiograms and IVUS imaging will be obtained.
Who Masked: Participant
Masking Description: The participant will be masked about which treatment strategy will be executed. Randomization will be done after diagnostic invasive pelvic angiography. The intervention procedure between both randomization groups is comparable, thus unmasking is difficult.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plain old balloon (POB) arm (Active Comparator): Balloon catheter used in the POB arm will be the "Medtronic" Euphora Rapid Exchange Balloon Dilatation Catheter, with diameters from 1.5 mm to 4.0 mm, and length from 6 to 30 mm,
  Interventions: Device: Plain old balloon angioplasty
- Drug-eluting balloon (DEB) arm (Experimental): The Selution SLR™ sirolimus-eluting balloon catheter system comprises of a semi-compliant polyamide balloon catheter with low tip profile coated with sirolimus drug (concentration: 1.00 μg/mm2 of balloon surface). Selution sustained limus release (SLR™) sirolimus-eluting balloon provides controlled and 90-day sustained release of sirolimus given its MicroReservoir technology made from biodegradable polymer intermixed with sirolimus. The balloon platform is the percutaneous transluminal coronary angioplasty (PTCA) rapid exchange catheter, with diameters from 2.0 to 4.5 mm and length from 15 to 30 mm.
  Interventions: Device: Selution SLR™ sirolimus-eluting balloon

INTERVENTIONS:
Device: Selution SLR™ sirolimus-eluting balloon — If the residual stenosis is ≤30% after initial plain old balloon angioplasty, the investigators will perform angioplasty with the Selution SLR catheter, inflated at nominal pressure for at least 120 seconds. After dilatation of the entire target-lesion, biplane angiograms and IVUS imaging will be obtained. Technical success is defined as residual diameter stenosis ≤30% and adequate distal run-off. Bail-out stenting will be performed if residual stenosis is >30%, either after plain old balloon angioplasty or angioplasty with Selution SLR. For lesions with residual stenosis >30% but not suitable for stenting, repeat angioplasty will be performed for at most twice.
  Arms: Drug-eluting balloon (DEB) arm
Device: Plain old balloon angioplasty — The investigators routinely start with a balloon catheter with a diameter ≥0.5 mm smaller than the reference vessel and ended with a balloon catheter with the size approximately equal to the reference vessel diameter. Three minutes after balloon predilation, the investigators will obtain an angiogram. If the residual stenosis is ≤30%, no further intervention will be performed in the plain old balloon (POB) group.
  Other Names: "Medtronic" Euphora Rapid Exchange Balloon Dilatation Catheter
  Arms: Plain old balloon (POB) arm

SUMMARY:
According to epidemiological surveys in various countries around the world, the prevalence of erectile dysfunction in men over the age of 40 is about 40%. Previous angiography studies have shown that nearly 70% of erectile dysfunction patients do have pelvic arterial stenosis. Our team leads the world in the use of percutaneous angioplasty combined with drug-eluting stents or paclitaxel-coated balloons to delineate the stenosis of the pelvic pudendal artery and penile artery The successful report of erectile dysfunction shows that the 12-month erectile function improvement rate is nearly 60%, and the vascular restenosis rate is also about 40% to 50%, obviously there is room for improvement. This study aims to observe the clinical efficacy, safety and lower restenosis rate of the newly developed "Selution SLR™ sirolimus drug sustained-release coated balloon" in patients with distal internal pudendal artery and penile artery stenosis complicated with erectile dysfunction . Compared with drug-eluting stents and paclitaxel drug-coated balloons, the Sirolimus drug-coated balloon has two advantages: one is that the clinical performance of sirolimus is much better than that of paclitaxel when used in drug-eluting stents; the other is that there is no indwelling stent in the Therefore, it can reduce the local stimulation of blood vessels and maintain the biological activity of blood vessels. Selution SLR™ sirolimus drug sustained-release coated balloon has obtained European Union approval for marketing, and has also been granted four Breakthrough Device Designation Status by the U.S. Food and Drug Administration (FDA): coronary artery disease, coronary artery disease In-stent restenosis, infra-knee artery disease, and arteriovenous canals.

DETAILED DESCRIPTION:
Study Design

1. Prospective, randomized, single-blinded, two-arm, single-center, first-in-man, proof-of-concept trial.
2. Safety and efficacy measures will be monitored and collected by the study physician/coordinator at hospital discharge, 2 weeks, 1, 3 (12 weeks), 6, and 8 (7-9, study end) months after the index procedure.
3. For patients developing binary restenosis at 12 weeks, angioplasty with Selution SLR drug-eluting balloon (in the drug-eluting balloon [DEB] arm) or plain old balloon (POB)(in the POB arm) will be performed thereafter and secondary patency will be evaluated 5 months later, the originally defined 8-month follow-up.

Target Population

1. Patient profile: Patients with erectile dysfunction according to International Index of Erectile Function-Erectile Function (IIEF-EF) score and distal internal pudendal and/or penile artery stenotic disease identified by pelvic computed tomography angiography (CTA) and confirmed by invasive angiography.
2. Inclusion criteria 2.1 Men ≥20 years of age with erectile dysfunction defined as an IIEF-EF score of ≤25 points; 2.2 The anatomical inclusion criteria, based on pelvic CT angiography, are luminal diameter stenosis of ≥50% in the distal internal pudendal and/or penile arteries with proximal reference vessel diameter of ≥1.5 mm and a target-lesion length of ≤40 mm.

Patients and Sites A total of 54 patients, with at least 54 evaluable lesions, from National Taiwan University Hospital will be enrolled in this trial. 1:2 randomization (18 and 36 in plain old balloon group and Selution group, respectively) will be performed. Pre-specified interim analyses for the primary efficacy outcome measure with an option to prematurely end the study will be conducted while 12, 20, 28, and 36 patients complete evaluation of the primary efficacy measure.

Primary Efficacy Endpoint CT angiographic binary restenosis (≥50% lumen diameter stenosis) at 12 weeks follow-up.

Primary Safety Endpoint The rate of major adverse events at 12 weeks after intervention, defined as procedure-related death, occurrence of perineal hematoma, gangrene or necrosis (glans penis, penile shaft, scrotal, or anal), or the need for subsequent perineal, penile, or anal surgery (including target-lesion or vessel revascularization or arterial embolization procedures).

Secondary Endpoints

1. Invasive angiographic binary restenosis (≥50% lumen diameter stenosis) at 8 (7-9) months follow-up;
2. CT angiographic binary restenosis (≥50% lumen diameter stenosis) at 8 (7-9) months follow-up;
3. Intravascular ultrasound (IVUS)-based binary restenosis (≥50% averaged lumen diameter stenosis) at follow-up;
4. Peak systolic velocity of treated-side cavernosal artery of >35 cm/sec by penile duplex ultrasonography at 12 weeks;
5. Technical success defined as residual diameter stenosis of ≤30% with adequate distal run-off (TIMI 3 flow) by invasive angiography 3 minutes after angioplasty with Selution SLR;
6. Change of IIEF-EF score at 1, 3, 6, and end of follow-up;
7. Clinical success defined as change of IIEF-EF score from baseline by ≥4 points or IIEF-EF ≥26 at 1, 3, 6, and end of follow-up;
8. Clinical worsening defined as decrease in IIEF-EF score from baseline by ≥4 points at 1, 3, 6, and end of follow-up;
9. Changes of invasive angiographic and IVUS parameters, including diameter, diameter stenosis, and late loss between 8 months and baseline;
10. Changes of CT angiographic parameters, including diameter, diameter stenosis, and late loss between 8 months and baseline;
11. Changes of penile duplex ultrasonographic parameters (peak systolic flow, RI) between follow-up and baseline;
12. The rates of major adverse events, defined as procedure-related death, occurrence of perineal hematoma, gangrene or necrosis (glans penis, penile shaft, scrotal, or anal), or the need for subsequent perineal, penile, or anal surgery (including target-lesion or vessel revascularization or arterial embolization procedures), at 1, 3 months, 6 months, and end of follow-up.

Statistical Considerations

1. Sample size estimation: Assuming a binary restenosis rate of 8% with Selution SLR sirolimus-eluting balloon versus a historical restenosis rate of 40% in patients treated with plain old balloon in our PERFECT registry, a minimum of 54 evaluable lesions in 54 patients with a 1:2 randomization ratio (18 and 36 in plain old balloon group and Selution group, respectively) was considered necessary to have a statistical power of 80% and a 2-sided p<0.05 to detect a treatment difference in binary restenosis. Pre-specified interim analyses for the primary efficacy outcome measure with an option to prematurely end the study will be conducted while 12, 20, 28, and 36 patients complete evaluation of the primary efficacy measure.
2. Statistical analysis This prospective, randomized, single-blinded (patient), two-arm, single-center, superiority study is a feasibility trial designed to provide preliminary observations and generate hypotheses for future studies. Continuous variables will be presented as means with standard deviations (SDs). Categorical variables will be presented as counts and percentages. Statistical comparisons between treatment groups will be made using t tests for continuous variables and χ² or Fisher's exact tests for categorical variables. Within each treatment group, paired t tests will be used to compare changes in continuous variables from baseline to follow-up.

Inclusion Criteria

1. Men ≥20 years of age with erectile dysfunction defined as an IIEF-EF score of ≤25 points;
2. The anatomical inclusion criteria, based on pelvic CT angiography, are luminal diameter stenosis of ≥50% in the distal internal pudendal and/or penile arteries with proximal reference vessel diameter of ≥1.5 mm and a target-lesion length of ≤40 mm;

Exclusion Criteria

1. The presence of diameter stenosis of ≥70% in the ipsilateral internal iliac artery, anterior division of internal iliac artery, and/or proximal internal pudendal artery, which could not be successfully treated by angioplasty and stenting;
2. Any non-vascular cause of erectile dysfunction (i.e., pelvic irradiation, pelvic trauma, Peyronie's disease, etc.), which is deemed irreversible by urologist;
3. Untreated hypogonadism (serum total testosterone <2.5 ng/ml) within 28 days before enrollment;
4. Isolated penile veno-occlusive dysfunction (venous leak) by duplex ultrasonography with right or left cavernosal artery end-diastolic velocity >10 cm/s, peak systolic velocity >40 cm/s, and resistance index (RI) <0.75;
5. Acute coronary syndrome, stroke, or life-threatening arrhythmia within 3 months before enrollment;
6. Poorly controlled diabetes mellitus with glycosylated hemoglobin levels >9%;
7. Serum creatinine levels >3.0 mg/dl;
8. Bleeding diathesis precluding the use of antiplatelets or anticoagulants or known hypercoagulopathy;
9. Any malignancy or debilitating disease with life expectancy of fewer than 12 months;
10. Known intolerance to contrast agents, aspirin, heparin, all P2Y12 inhibitors, or sirolimus.

Procedure All patients will be admitted one day prior to the procedure and receive aspirin (100 mg daily) and clopidogrel (75 mg daily and 300 mg loading one day before intervention) 24 h prior to the procedure. Selective angiography and internal pudendal/penile artery interventions will be performed on the second day of hospitalization. All procedures will be done percutaneously by an over-the-bifurcation (for the contralateral lesions) or a retrograde (for the ipsilateral lesions) approach via a single femoral vascular access with the use of a 6-French sheath. The investigators routinely engage the proximal internal pudendal artery by using a 5-French diagnostic/guiding catheter and obtain the selective angiograms following intraarterial administration of 150-200 microg of nitroglycerin to achieve maximal vasodilatation. Use of any phosphodiesterase-5 inhibitor within 72 hours of the procedure will be prohibited.

Patients will proceed with investigational intervention if their quantitative angiographic results fulfilled the following angiographic inclusion criteria: 1) luminal diameter stenosis of ≥50% in the distal internal pudendal and/or penile arteries, 2) a target-lesion proximal reference vessel diameter ≥1.5 mm, and 3) a target-lesion length ≤40 mm. Patients will be excluded if there is ≥70% stenosis in the ipsilateral ilio-pudendal-penile arterial system proximal to the distal internal pudendal artery and not amenable to interventional therapy.

After confirmation of angiographic eligibility, patients will receive 8,000 U of heparin to maintain an activated clotting time ≥250 s. Selective engagement of the internal pudendal artery will be performed with an appropriate-shaped 5-French guiding catheter. A 0.014-inch steerable guidewire will be advanced across the stenosis and IVUS and standard interventional techniques will be applied to the lesion. In order to prevent inadvertent dissection during predilation, the investigators routinely start with a balloon catheter with a diameter ≥0.5 mm smaller than the reference vessel and ended with a balloon catheter with the size approximately equal to the reference vessel diameter. Three minutes after balloon predilation, the investigators will obtain an angiogram. Randomization will take place before angioplasty. If the residual stenosis is ≤30%, no further intervention will be performed in the plain old balloon (POB) group. While in the drug-eluting balloon (DEB) group, the investigators will perform angioplasty with the Selution SLR catheter, inflated at nominal pressure for at least 120 seconds. After dilatation of the entire target-lesion, biplane angiograms and IVUS imaging will be obtained. Technical success is defined as residual diameter stenosis ≤30% and adequate distal run-off. Bail-out stenting will be performed if residual stenosis is >30%, either after plain old balloon angioplasty or angioplasty with Selution SLR. For lesions with residual stenosis >30% but not suitable for stenting, repeat angioplasty will be performed for at most twice.

After intervention, patients will be discharged in the morning of the third day of hospitalization. Post-procedural antiplatelet therapy include aspirin (100 mg daily) indefinitely and clopidogrel (75 mg daily) for a minimum of 3 months.

Patient Follow-up

1. Safety and efficacy measures will be monitored and collected by the study physician/coordinator at hospital discharge, 2 weeks, 1, 3, 6, and 8 (7-9, study end) months after the index procedure. Participants will be encouraged to contact the study physician/coordinator directly by phone whenever the participants feel any discomfort, no matter it is related to the procedure or not.
2. For patients developing binary restenosis at 12 weeks, angioplasty with plain old balloon (in the POB arm) or Selution SLR drug-eluting balloon (in the DEB arm) will be performed thereafter and secondary patency will be evaluated 5 months later, the originally defined 8-month follow-up.
3. For patients developing binary restenosis at 8 months, angioplasty with Selution SLR drug-eluting balloon will be performed. All these patients will be followed for additional 6 months.

Safety Monitoring Safety events including procedure-related death, occurrence of perineal hematoma, gangrene or necrosis (glans penis, penile shaft, scrotal, or anal), or the need for subsequent perineal, penile, or anal surgery (including target-lesion or vessel revascularization or arterial embolization procedures) will be collected by the study physician/coordinator at 1, 3, 6 months, and study end after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥20 years of age with erectile dysfunction defined as an IIEF-EF score of ≤25 points;
2. Inadequate response to any dosage of phosphodiesterase 5 inhibitor (PDE5i) for more than 6 months before enrollment (either chronic or on-demanding).
3. Hemodynamic conditions stable (systolic BP > 100 mmHg, heart rate 40-100/min).
4. The anatomical inclusion criteria, based on pelvic CT angiography, are luminal diameter stenosis of ≥50% in the distal internal pudendal and/or penile arteries with proximal reference vessel diameter of ≥1.5 mm and a target-lesion length of ≤40 mm;

Exclusion Criteria:

1. The presence of diameter stenosis of ≥70% in the ipsilateral internal iliac artery, anterior division of internal iliac artery, and/or proximal internal pudendal artery, which could not be successfully treated by angioplasty and stenting;
2. Any non-vascular cause of erectile dysfunction (i.e., pelvic irradiation, pelvic trauma, Peyronie's disease, etc.), which is deemed irreversible by urologist;
3. Untreated hypogonadism (serum total testosterone <2.5 ng/ml) within 28 days before enrollment;
4. Isolated penile veno-occlusive dysfunction (venous leak) by duplex ultrasonography with right or left cavernosal artery end-diastolic velocity >10 cm/s, peak systolic velocity >40 cm/s, and resistance index (RI) <0.75;
5. Acute coronary syndrome, stroke, or life-threatening arrhythmia within 3 months before enrollment;
6. Poorly controlled diabetes mellitus with glycosylated hemoglobin levels >9%;
7. Patient on dialysis or has known renal insufficiency (serum creatinine > 2.5 mg/dl, or estimated Glomerular Filtration Rate <30 ml/min/1.732);
8. Serum creatinine levels >3.0 mg/dl;
9. Bleeding diathesis (like active peptic ulcer, active bleeding, etc.) precluding the use of antiplatelets or anticoagulants or known hypercoagulopathy;
10. Any malignancy or debilitating disease with life expectancy of fewer than 12 months;
11. Known intolerance to contrast agents, aspirin, heparin, all P2Y12 inhibitors, or sirolimus.
12. Severe hepatic insufficiency;

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 12 weeks
  CT angiographic binary restenosis (≥50% lumen diameter stenosis) at 12 weeks follow-up.
Primary safety endpoint | 12 weeks
  The rate of major adverse events at 12 weeks after intervention, defined as procedure-related death, occurrence of perineal hematoma, gangrene or necrosis (glans penis, penile shaft, scrotal, or anal), or the need for subsequent perineal, penile, or anal surgery (including target-lesion or vessel revascularization or arterial embolization procedures).

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Tzung-Dau Wang, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang TD, Lee CK, Chia YC, Tsoi K, Buranakitjaroen P, Chen CH, Cheng HM, Tay JC, Teo BW, Turana Y, Sogunuru GP, Wang JG, Kario K; HOPE Asia Network. Hypertension and erectile dysfunction: The role of endovascular therapy in Asia. J Clin Hypertens (Greenwich). 2021 Mar;23(3):481-488. doi: 10.1111/jch.14123. Epub 2020 Dec 14. PMID 33314715
- [Result] Wang TD, Lee WJ, Yang SC, Lin PC, Tai HC, Liu SP, Huang CH, Chen WJ, Chen MF, Hsieh JT. Clinical and Imaging Outcomes up to 1 Year Following Balloon Angioplasty for Isolated Penile Artery Stenoses in Patients With Erectile Dysfunction: The PERFECT-2 Study. J Endovasc Ther. 2016 Dec;23(6):867-877. doi: 10.1177/1526602816669337. Epub 2016 Sep 14. PMID 27629440
- [Result] Wang TD, Lee WJ, Yang SC, Lin PC, Tai HC, Hsieh JT, Liu SP, Huang CH, Chen WJ, Chen MF. Safety and six-month durability of angioplasty for isolated penile artery stenoses in patients with erectile dysfunction: a first-in-man study. EuroIntervention. 2014 May;10(1):147-56. doi: 10.4244/EIJV10I1A23. PMID 24832642
- [Result] Wang TD. Commentary: Angioplasty of Internal Pudendal and Penile Arteries for Arteriogenic Erectile Dysfunction: Reassuring, but the Jury Is Still Out. J Endovasc Ther. 2018 Dec;25(6):716-718. doi: 10.1177/1526602818807774. Epub 2018 Oct 22. No abstract available. PMID 30343618